CLINICAL TRIAL: NCT04482426
Title: Correlates of Electrophysiological Activities in Different Pelvic Floor Muscle Groups and Female Pelvic Floor Function
Acronym: PFMF
Status: Completed | Type: Observational
Sponsor: Cathay General Hospital (Other)
Responsible Party: Principal Investigator, Wen-Chen Huang, Professor, Cathay General Hospital
Other Study IDs: CGH-P102071
Record Dates: First submitted 2020-07-19; First posted 2020-07-22 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Pelvic Floor

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

SUMMARY:
The study aimed to explore and quantify functional and electrical activities in different pelvic floor muscle groups, to differentiate the electrophysiological role in different pelvic floor muscle groups relating to pelvic floor dysfunction or disorders, and further to develop treatment strategies for different pelvic floor muscle groups in different female pelvic disorders.

DETAILED DESCRIPTION:
Female pelvic floor disorders including sexual dysfunction, urinary incontinence, fecal incontinence, and pelvic organ prolapse are relating to the function of pelvic floor structures. Essential components responsible for pelvic floor function include bony, muscular, and fascial structures of the pelvis. Among above components, pelvic floor muscles, either the superficial or deep group, are considered crucial in maintaining the morphology and functional integrity of the pelvic floor.

Inspection and digital examination incorporating Oxford grading system during pelvic examinations are the most convenient and commonly methods applied to evaluate the function of pelvic floor muscles. Nevertheless, both methods cannot provide quantitative information of pelvic floor muscle contraction. With the introduction of pelvic floor manometry and electrophysiological testing, quantification of pelvic floor muscle contractions can be expected.

The study aimed to explore and quantify functional and electrical activities in different pelvic floor muscle groups, to differentiate the electrophysiological role in different pelvic floor muscle groups relating to pelvic floor dysfunction or disorders, and further to develop treatment strategies for different pelvic floor muscle groups in different female pelvic disorders.

ELIGIBILITY:
Inclusion Criteria:

* Women with pelvic floor dysfuntion

Exclusion Criteria:

* Pregnant women
* Women with histories of diabetes, cerebrovascular diseases, neurological diseases, degenerative muscular diseases, or autoimmune connective tissue diseases。

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with pelvic floor dysfunction
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2014-07-25; Primary Completion 2015-08-29 (Actual); Study Completion 2017-08-11 (Actual)

PRIMARY OUTCOMES:
Contraction of pelvic floor muscle | Baseline
  Chart review